CLINICAL TRIAL: NCT00146159
Title: A Double-Blind, Three-Armed, Randomized Phase-III-Study, to Compare the Efficacy, Tolerability and Safety of Three Doses of Mitoxantrone in the Treatment of Patients With Secondary Progressive Multiple Sclerosis
Brief Title: Study Evaluating Mitoxantrone in Multiple Sclerosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Clinical Trials Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0906E-100925
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Mitoxantrone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): 1st group: 12 mg Mitoxantrone/m²
  Interventions: Drug: Mitoxantrone
- 2 (Experimental): 2nd group: 9mg Mitoxantrone/m²
  Interventions: Drug: Mitoxantrone
- 3 (Experimental): 3rd group: 5mg Mitoxantrone/m²
  Interventions: Drug: Mitoxantrone

INTERVENTIONS:
Drug: Mitoxantrone — dosage

SUMMARY:
The purpose of this study is to show the dose-response relationship of three doses of mitoxantrone with regard to efficacy in patients with secondary progressive multiple sclerosis and to show the safety and tolerability of mitoxantrone in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Secondary progressive MS in an active stage
* EDSS between 3 and 6

Exclusion Criteria:

* Benign or primary progressive MS
* Patients with cardiac risk factors
* Patients who have already received mitoxantrone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 336 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
3 clinical measures combined in a multivariate analysis: confirmed Expanded Disability Status Scale(EDSS) | 3 years
deterioration, change of ambulation index, time to first relapse requiring corticoid treatment | 3 years

SECONDARY OUTCOMES:
derivations of EDSS and relapses; MRI (baseline, 2 years) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (6):
- Germany (6):
  - Berg
  - Berlin
  - Düsseldorf
  - Giessen
  - Marburg
  - Wiesbaden